CLINICAL TRIAL: NCT05858333
Title: Pregnancy Outcome of Extended Culture of Day 3 to Day 5 Frozen Thawed Day 3 Embryos Versus Day 5 Frozen-Thawed Embryos
Brief Title: Extended Culture of Day 3 to Day 5 Frozen Thawed Day 3 Embryos Versus Day 5 Frozen-Thawed Embryos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Sennara, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: vitrification of embryos
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: (day 5 group) (No Intervention): Women will undergo ICSI, and verification-thawed blastocysts will be transferred after 5 days of ovulation (60cases).
- Group 2: (day 3-5 group) (Experimental): Women will undergo ICSI, who had cryopreserved embryos on day 3 then thawed and embryos will be allowed for extended cultured for 2 additional days and then will be transferred as blastocysts after 5 days of ovulation (60 cases).
  Interventions: Other: Extended culture for Group 2: (day 3-5 group)

INTERVENTIONS:
Other: Extended culture for Group 2: (day 3-5 group) — To investigate thawing day three embryos and culturing them to be transferred as blastocyst that will improve pregnancy rate when compared to transfer thawed frozen blastocyst.
  Arms: Group 2: (day 3-5 group)

SUMMARY:
Cryopreservation of embryos and oocytes has become routine in assisted reproduction technology (ART). Live birth rates following frozen embryo transfers have increased significantly. Data show that cryopreservation has significant improved survival rates and cumulative pregnancy rates, as well as the safety of ART . Embryo cryopreservation has become a cornerstone in ART. With improved vitrification techniques. Frozen embryos transfer (FET) shows equal or even higher implantation and pregnancy rates than do fresh embryo transfers ART Previous studies show equal or even superior outcomes regarding pregnancy and live birth rates with frozen versus fresh embryo transfer Cryopreserve all embryos have increased substantially in recent years, and according to the recent trend of a freeze-all strategy. This study aims to answer a clinical question encountered in daily practice regarding at what stage embryos should be frozen.

DETAILED DESCRIPTION:
Cryopreservation of embryos and oocytes has become routine in assisted reproduction technology (ART). Live birth rates following frozen embryo transfers have increased significantly. Data show that cryopreservation has significant improved survival rates and cumulative pregnancy rates, as well as the safety of ART. Embryo cryopreservation has become a cornerstone in ART. With improved vitrification techniques. Frozen embryos transfer (FET) shows equal or even higher implantation and pregnancy rates than do fresh embryo transfers ART .

Previous studies show equal or even superior outcomes regarding pregnancy and live birth rates with frozen versus fresh embryo transfer .

Cryopreservation has several advantages. It maintains supernumerary embryos not used for fresh transfer; allows single-embryo transfer, thus reducing multiple gestations; enables a freeze-all strategy to prevent ovarian hyper stimulation syndrome; is useful for social or medical fertility preservation; and allows embryo biopsy for preimplantation genetic testing, luteal phase stimulation, and dual stimulation protocols .

A recent trend is to perform blastocyst fresh/frozen single-embryo transfers. The advantages include exposing the embryo to a more natural uterine environment. Also, by extending the duration of culture, embryo self-selection will occur and may enable the highest chance of implantation . Due to a potential damage to the expanded blastocyst during vitrification procedure, an emerging clinical question is whether cryopreserving cleavage stage embryos, then thawing and culturing to blastocysts will achieve better outcomes, as compared to transfer of a thawed blastocyst .

The most recent study demonstrated that thawing cleavage embryos, then culturing and transferring them as blastocysts, yields improved pregnancy rates and perinatal outcomes compared to thawed blastocyst embryo transfers . Cryopreserve all embryos have increased substantially in recent years, and according to the recent trend of a freeze-all strategy. This study aims to answer a clinical question encountered in daily practice regarding at what stage embryos should be frozen.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with history of primary or secondary infertility.
2. Age ≤ 38 years.
3. Female patients having more than 4 vitrified embryos.
4. BMI less than 30 kg/m².
5. Good quality of embryos

Exclusion Criteria:

1. Severe male factor infertility.
2. Recurrent implantation failure.
3. Females with uterine Congenital anomalies.
4. Bad quality of embryos.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women who will transfer frozen embryos
Enrollment: 132 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-09-17 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
To increase the pregnancy rate of cases undergoes to ICSI. | 16 months
  Pregnancy rates will be determined in each of the two groups and compared to each other in three stages in clinical pregnancy, ongoing pregnancy and live pregnancy rates.

CONTACTS AND LOCATIONS:
Locations (1):
- International Islamic Center for Population Studies and Researches (IICPSR) - Al-Azhar University, Cairo, Al-Azhar University, Al-Darrasah, Egypt

REFERENCES:
- [Background] Boyard J, Reignier A, Chtourou S, Lefebvre T, Barriere P, Freour T. Should artificial shrinkage be performed prior to blastocyst vitrification? A systematic review of the literature and meta-analysis. Hum Fertil (Camb). 2022 Feb;25(1):24-32. doi: 10.1080/14647273.2019.1701205. Epub 2020 Jan 24. PMID 31973647
- [Background] Gardner DK, Lane M, Stevens J, Schlenker T, Schoolcraft WB. Blastocyst score affects implantation and pregnancy outcome: towards a single blastocyst transfer. Fertil Steril. 2000 Jun;73(6):1155-8. doi: 10.1016/s0015-0282(00)00518-5. PMID 10856474
- [Background] Martins WP, Nastri CO, Rienzi L, van der Poel SZ, Gracia C, Racowsky C. Blastocyst vs cleavage-stage embryo transfer: systematic review and meta-analysis of reproductive outcomes. Ultrasound Obstet Gynecol. 2017 May;49(5):583-591. doi: 10.1002/uog.17327. Epub 2017 Apr 10. PMID 27731533
- [Background] Nagy ZP, Shapiro D, Chang CC. Vitrification of the human embryo: a more efficient and safer in vitro fertilization treatment. Fertil Steril. 2020 Feb;113(2):241-247. doi: 10.1016/j.fertnstert.2019.12.009. PMID 32106970
- [Background] Ozgur K, Berkkanoglu M, Bulut H, Isikli A, Coetzee K. Higher clinical pregnancy rates from frozen-thawed blastocyst transfers compared to fresh blastocyst transfers: a retrospective matched-cohort study. J Assist Reprod Genet. 2015 Oct;32(10):1483-90. doi: 10.1007/s10815-015-0576-1. Epub 2015 Sep 23. PMID 26400506
- [Background] Rahav-Koren R, Inbar S, Miller N, Wiser A, Yagur Y, Berkowitz C, Farladansky-Gershnabel S, Shulman A, Berkowitz A. Thawing day 3 embryos and culturing to day 5 may be a better method for frozen embryo transfer. J Assist Reprod Genet. 2021 Nov;38(11):2941-2946. doi: 10.1007/s10815-021-02321-y. Epub 2021 Sep 22. PMID 34549329
- [Background] Roque M, Haahr T, Geber S, Esteves SC, Humaidan P. Fresh versus elective frozen embryo transfer in IVF/ICSI cycles: a systematic review and meta-analysis of reproductive outcomes. Hum Reprod Update. 2019 Jan 1;25(1):2-14. doi: 10.1093/humupd/dmy033. PMID 30388233
- [Background] Van Landuyt L, Polyzos NP, De Munck N, Blockeel C, Van de Velde H, Verheyen G. A prospective randomized controlled trial investigating the effect of artificial shrinkage (collapse) on the implantation potential of vitrified blastocysts. Hum Reprod. 2015 Nov;30(11):2509-18. doi: 10.1093/humrep/dev218. Epub 2015 Sep 12. PMID 26364080
- [Background] Wang A, Santistevan A, Hunter Cohn K, Copperman A, Nulsen J, Miller BT, Widra E, Westphal LM, Yurttas Beim P. Freeze-only versus fresh embryo transfer in a multicenter matched cohort study: contribution of progesterone and maternal age to success rates. Fertil Steril. 2017 Aug;108(2):254-261.e4. doi: 10.1016/j.fertnstert.2017.05.007. Epub 2017 Jun 1. PMID 28579411